CLINICAL TRIAL: NCT05649865
Title: Analysis of HPV DNA in Plasma in Patients With HPV-positive Oropharyngeal Squamous Cell Carcinoma - a Prospective Study of HPV DNA Levels for Treatment Response and Surveillance
Brief Title: Monitoring and Early Response Evaluation Using HPV DNA - A Study on Patients With HPV-positive Throat Cancer (MER-HPV)
Acronym: MER-HPV
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-04539-01
Record Dates: First submitted 2022-11-17; First posted 2022-12-14 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Oropharynx Squamous Cell Carcinoma
Keywords: Human papilloma virus; circulating HPV DNA
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — HPV DNA will be analyzed from the primary tumour tissue and circulating tumour HPV DNA will be analyzed in plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with HPV-positive OPC: Patients with HPV-positive OPC. They will provide blood samples before during and after treatment to evaluate treatment response and for early detection of recurrence
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Blood samples for analysis of circulating tumour HPVDNA

SUMMARY:
The goal of this clinical trial is to determine the value of circulating tumour HPV DNA (human papilloma virus DNA found in the blood) at diagnosis, during treatment, and in the follow-up of patients diagnosed and treated for throat cancer caused by HPV.

The main question to answer is if the presence of HPV DNA in the blood one month after the treatment is useful in detecting remaining tumour or relapse within two years after treatment.

The participants will be asked to provide blood tests:

1. before treatment
2. weekly during the treatment
3. on all scheduled follow-up appointments
4. on all unplanned appointments where a relapse is suspected

DETAILED DESCRIPTION:
Background:

There is a yearly increase in the incidence of oropharyngeal carcinoma (OPC) of appr. 5% in Sweden, predominantly in males. More than 80% of the tumours are HPV (human papilloma virus)-positive. For that reason, measuring circulating tumour HPV DNA (ctHPVDNA) in plasma as a marker of treatment response and as an adjunct in surveillance has become an appealing possibility.

In Sweden, patients intended for curative treatment for OPC are usually treated with (chemo)radiotherapy (c)RT. A small proportion is subjected to surgery with or without adjuvant radiation. The gold standard for treatment evaluation after definitive (c)RT is a positron emission tomography-computed tomography (PET-CT) performed 12 weeks after (c)RT completion. The PET-CT result is most important to determine the need for neck dissection in patients with node-positive disease at diagnosis.

According to previous publications on the subject of ctHPVDNA, there are the following reasons to further explore the value of ctHPVDNA in routine clinical practice in patients with HPV-positive OPC:

1. ctHPVDNA might limit or almost distinguish the issue with PET-CT results assessed as equivocal treatment evaluation response. A combination of the PET-CT result and ctHPVDNA analysis seems to increase the accuracy.
2. ctHPVDNA has a great potential to detect recurrences before subjective symptoms occur and before it becomes apparent on clinical examination. Early detection of distant metastases in this group of patients might be valuable, since they have the potential for prolonged overall survival after salvage therapy compared to HPV-negative patients. And detection of a small tumour burden might improve survival further.
3. An accurate detection of recurrences with ctHPVDNA in plasma might lead to a discussion of reducing scheduled follow-up appointments and following the patients with plasma samples instead.

All patients with biopsy proven OPC referred to the Dept. of Otorhinolaryngology-Head and Neck Surgery (ORL-HNS), Skåne University Hospital and planned for definitive treatment as decided at the Multidisciplinary Tumour Board (MDT) will be invited to participate. Only patients with an HPV-positive tumour are eligible for inclusion.

Sample size calculated for the primary end-point:

A sensitivity of 65% for detectable ctHPVDNA at one month was decided to be of clinical value for predicting residual or recurrent tumour within two years after treatment completion. 15% of the patients were estimated not to reach complete remission after primary (c)RT or suffer from recurrence during a two-year follow-up period. Accordingly, a sensitivity of at least 65% requires a sample size of 150 patients with a power of 80%. Clopper-Pearson was used to calculate binomial CI of 95%.

The expectation is that 2/3 of the patients will be male, according to the epidemiology of OPC in Sweden.

Procedure and ctHPVDNA samples during treatment:

Patients will receive oral and written information of the study at their first visit at the Dept. of Oncology/Dept. of ORL.

Informed consent will be collected at the Dept. of Oncology. The patients will be followed for five years. The study will be closed when the last included patient has been followed for three years after treatment.

Plasma samples for ctHPVDNA analysis will be collected before (c)RT start or before surgery.

Weekly samples, i.e., seven, are planned during the course of radiotherapy (RT).

In surgically treated patients, two samples will be collected. The first at postoperative day 1 and the second on postoperative day 3. If the patient is recommended adjuvant (c)RT weekly samples will be collected as described above.

Treatment evaluation:

For treatment evaluation and surveillance, plasma ctHPVDNA will be analysed one month after treatment completion and then every three months during the first two years and every six months year two-five after treatment i.e, at the same time as the scheduled follow-up appointments according to the national guidelines.

For treatment evaluation at three months after (C)RT, the levels of ctHPVDNA will be taken into consideration as additive information to PET CT for the evaluation of treatment response. If the PET-CT is assessed as NI-RADS 1-2 but the ctHPVDNA level is increasing compared with the level at the end of treatment, a new test will be performed two weeks later to decide whether additional work-up is recommended. Patients with a complete PET CT response (i.e., NI-RADS 1-2) and non-detectable levels of ctHPVDNA will proceed directly to the follow-up regimen. Additional work-up e.g., timing of repeat imaging or other further examinations will be at the discretion of the MDT.

For treatment evaluation at three months after primary surgery increasing levels of ctHPVDNA will prompt a confirming test two weeks later to decide whether work-up is indicated. If the patient has decreasing levels of ctHPVDNA the participant will proceed to the follow-up regimen.

During follow-up (i.e., from six months and onwards), a positive ctHPVDNA test will be confirmed with a new test two weeks later. If a confirmation of detectable ctHPVDNA levels is achieved, a recurrence work-up will be initiated, including PET CT and further examinations at the discretion of the MDT and scheduled accordingly.

Baseline and follow-up data:

Baseline data includes age, sex, smoking status, any previous head and neck cancer (HNC), date of diagnosis, primary tumour subsite, TNM classification/stage, p16-status, HPV subtype in primary tumour, levels of ctHPVDNA before treatment.

Follow-up data includes received treatment, clinical response three months after treatment, clinical status at the scheduled clinical reviews as well as additional reviews for clinical suspicion of recurrence, PET-CT response at 12 weeks after treatment according to NI-RADS, results of any additional imaging related to HNC, ctHPVDNA i plasma, reasons for aborting treatment and or terminate scheduled reviews, any recurrence, date of death, cause of death, alive with or without disease at five years of follow-up or when the study is closed.

Recurrence:

If the patient is diagnosed with a residual tumour or recurrence planned for curative intent the plasma sample scheme for ctHPVDNA will be recommenced. If palliative treatment is started after a recurrence no further plasma samples will be collected. A recurrence is diagnosed when a positive cytology or biopsy confirms cancer or if progressive disease is verified on imaging. The date when the cytology or biopsy was performed will serve as the date of recurrence. The first suspicion of a radiology defined recurrence will serve as the date of recurrence if the patient is deemed unfit for confirmation with cytology or biopsy.

Method for HPV-DNA analysis:

HPV-DNA type identification and quantification from the primary tumour and ctHPV-DNA-quantification in plasma, from each patient, are performed with Luminex and ddPCR, respectively. Luminex is performed at the Dept. of Microbiology, and digital droplet polymerase chain reaction (ddPCR) at the Center for Molecular Diagnostics (CMD), Lund.

Primary tumour:

Tumour sample, in formalin, is sent to Dept. of Microbiology, Lund. Then sections from formalin fixed paraffin-embedded (FFPE) tumour-tissue are delivered to Dept. of Microbiology. DNA from formalin fixed paraffin-embedded (FFPE) tissue will be extracted according to established standard methods at Dept. of Microbiology. HPV type will be determined by PCR followed by Luminex-based genotyping. If the tumour is HPV-positive, quantitative viral load (number of HPV copies per human cell) will be determined by ddPCR containing primers and probes specific for the HPV type demonstrated in the tumour.

Plasma:

Blood sample 8.5mL, is collected in vacutainer tube (BD ACD-A tube) and sent to Dept. of Microbiology, Lund. Plasma is separated by centrifugation at 1700 xRPM at Dept. of Microbiology. Then ctDNA is extracted from the plasma automatically by a QIAsymphony-robot using the DSP Circulating DNA Kit (Qiagen) (3 mL input 60 uL output). HPV type specific ddPCR, with primers and probes specific for the HPV type demonstrated in the tumour, will be performed to determine viral load (number of HPV copies per mL plasma).

Data monitoring:

The study is partly exploratory and partly performed as an evaluation of ctHPVDNA as a way of monitoring disease status. No adverse effects are expected. There is no monitoring committee or stopping guidelines. An interim analysis will be performed after the inclusion of 50 patients to secure the inclusion pace and evaluate unexpected problems. Internal validation will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Only patients with an HPV-positive primary tumour will eventually be eligible for inclusion.

   Non-detectable ctHPVDNA at diagnosis will not be a reason for exclusion.
2. Age >18 years.
3. Able to give informed consent.
4. The patient will be treated with curative intent.

Exclusion Criteria:

Patients with a short life expectancy, psychiatric or addictive disorders, or other medical conditions which might impair patient compliance may be excluded at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients in the Southern Health Care Region of Sweden, referred to Skane University Hospital, Lund, Sweden for curative treatment of HPV-positive oropharyngeal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of detectable ctHPVDNA one month after (c)RT completion | From inclusion to two years after treatment
  To determine if detectable ctHPVDNA one month post (C)RT is useful to detect residual or recurrent tumours diagnosed within two years.

OTHER OUTCOMES:
The correlation of ctHPVDNA with stage/tumour burden. | 2 weeks after inclusion
  Analyse the possible correlation of ctHPVDNA with stage/tumour burden.
The correlation of ctHPVDNA titer decay during treatment with residual tumour. | From inclusion to 3 months after the end of treatment
  Explore ctHPVDNA titer decay during the course of RT and surgery its relation to residual tumour evaluated at six months post treatment.
The correlation of ctHPVDNA levels with PET response and pathology reports for treatment evaluation. | From inclusion to 6 months after the end of treatment
  Determine the additive value of ctHPVDNA in addition to PET response for treatment evaluation after (C)RT. The assessment will be performed at six months post treatment.
The negative predictive value (NPV) and positive predictive value (PPV) of ctHPVDNA in relation to locoregional and and metastatic recurrence. | From inclusion to three years after the end of treatment
  Define the NPV and PPV of ctHPVDNA in relation to locoregional and metastatic recurrence diagnosed within three years after treatment completion.
The correlation of ctHPVDNA with clinical examinations post treatment. | From inclusion to three years after the end of treatment
  Assess the additive value of ctHPVDNA to clinical examinations post treatment.
Analyse the prognostic value of ctHPVDNA levels at diagnosis. | From inclusion to three years after the end of treatment
  The correlation of ctHPVDNA levels at diagnosis with progression free and overall survival.
The correlation of smoking on ctHPVDNA dynamics and treatment outcome. | From inclusion to three years after the end of treatment
  Define the influence of smoking on ctHPVDNA dynamics and treatment outcome.
Progression free and overall survival endpoints compared with a matched cohort from the Swedish Head and Neck Cancer Register (SweHNCR). | From inclusion to three years after the end of treatment
  Compare progression free and overall survival endpoints with a matched cohort from the Swedish Head and Neck Cancer Register (SweHNCR).

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Sjövall, MD,PhD, Principal Investigator — Dept. of clincial sciences, Lund University
Locations (1):
- Dept. of ORL-HNS, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammarstedt L, Lindquist D, Dahlstrand H, Romanitan M, Dahlgren LO, Joneberg J, Creson N, Lindholm J, Ye W, Dalianis T, Munck-Wikland E. Human papillomavirus as a risk factor for the increase in incidence of tonsillar cancer. Int J Cancer. 2006 Dec 1;119(11):2620-3. doi: 10.1002/ijc.22177. PMID 16991119
- [Background] Haring CT, Dermody SM, Yalamanchi P, Kang SY, Old MO, Chad Brenner J, Spector ME, Rocco JW. The future of circulating tumor DNA as a biomarker in HPV related oropharyngeal squamous cell carcinoma. Oral Oncol. 2022 Mar;126:105776. doi: 10.1016/j.oraloncology.2022.105776. Epub 2022 Feb 17. PMID 35183912
- [Background] Chera BS, Kumar S, Shen C, Amdur R, Dagan R, Green R, Goldman E, Weiss J, Grilley-Olson J, Patel S, Zanation A, Hackman T, Blumberg J, Patel S, Thorp B, Weissler M, Yarbrough W, Sheets N, Mendenhall W, Tan XM, Gupta GP. Plasma Circulating Tumor HPV DNA for the Surveillance of Cancer Recurrence in HPV-Associated Oropharyngeal Cancer. J Clin Oncol. 2020 Apr 1;38(10):1050-1058. doi: 10.1200/JCO.19.02444. Epub 2020 Feb 4. PMID 32017652
- [Background] Rutkowski TW, Mazurek AM, Snietura M, Hejduk B, Jedrzejewska M, Bobek-Billewicz B, d'Amico A, Piglowski W, Wygoda A, Skladowski K, Kolosza Z, Widlak P. Circulating HPV16 DNA may complement imaging assessment of early treatment efficacy in patients with HPV-positive oropharyngeal cancer. J Transl Med. 2020 Apr 15;18(1):167. doi: 10.1186/s12967-020-02330-y. PMID 32293457
- [Background] Tanaka H, Takemoto N, Horie M, Takai E, Fukusumi T, Suzuki M, Eguchi H, Komukai S, Tatsumi M, Isohashi F, Ogawa K, Yachida S, Inohara H. Circulating tumor HPV DNA complements PET-CT in guiding management after radiotherapy in HPV-related squamous cell carcinoma of the head and neck. Int J Cancer. 2021 Feb 15;148(4):995-1005. doi: 10.1002/ijc.33287. Epub 2020 Sep 30. PMID 32895945
- [Background] O'Boyle CJ, Siravegna G, Varmeh S, Queenan N, Michel A, Pang KCS, Stein J, Thierauf JC, Sadow PM, Faquin WC, Wang W, Deschler DG, Emerick KS, Varvares MA, Park JC, Clark JR, Chan AW, Busse PM, Corcoran RB, Wirth LJ, Lin DT, Iafrate AJ, Richmon JD, Faden DL. Cell-free human papillomavirus DNA kinetics after surgery for human papillomavirus-associated oropharyngeal cancer. Cancer. 2022 Jun 1;128(11):2193-2204. doi: 10.1002/cncr.34109. Epub 2022 Feb 9. PMID 35139236
- [Background] Routman DM, Kumar S, Chera BS, Jethwa KR, Van Abel KM, Frechette K, DeWees T, Golafshar M, Garcia JJ, Price DL, Kasperbauer JL, Patel SH, Neben-Wittich MA, Laack NL, Chintakuntlawar AV, Price KA, Liu MC, Foote RL, Moore EJ, Gupta GP, Ma DJ. Detectable Postoperative Circulating Tumor Human Papillomavirus DNA and Association with Recurrence in Patients With HPV-Associated Oropharyngeal Squamous Cell Carcinoma. Int J Radiat Oncol Biol Phys. 2022 Jul 1;113(3):530-538. doi: 10.1016/j.ijrobp.2022.02.012. Epub 2022 Feb 12. PMID 35157995